CLINICAL TRIAL: NCT03011827
Title: Transfusion Prediction Model in Orthotopic Liver Transplantation Based on Thromboelastometry: Prospective Validation Study.
Brief Title: Thromboelastometry in Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Annabel Blasi, Anesthesiologist, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATR100F
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Liver Transplant Disorder; Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective cohort (Experimental): Fibrinogen and/or platelet administration
  Interventions: Other: Fibrinogen and/or platelets administration

INTERVENTIONS:
Other: Fibrinogen and/or platelets administration — Fibrinogen and/or platelets administration to maintain clot amplitude at 10 minutes of the thromboelastometry between 35-40 mm along liver transplant procedure

SUMMARY:
Thromboelastometry better assess coagulation than standard coagulation test in patients undergoing ortothopic liver transplantation. In a post-hoc analysis from a randomized study recently conducted by our group, presurgical values of MA10 Extem < 35 mm are highly predictive of RBC administration , with no further improvement over MA10 Extem >40 mm ; suggesting that MA10 Extem between 35-40 would be the optimal range to manage blood product administration. The aim of the study is to validate this result in a prospective cohort of patients submitted to ortothopic liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Presurgical hemoglobin < 13 d/L and clot firmness at 10 minutes Extem < 35 mm

Exclusion Criteria:

* Previous thrombosis
* Antithrombotic treatment
* No consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Red blood cell transfusion | until 24h after liver transplant

SECONDARY OUTCOMES:
Thrombosis | 28 days after liver transplant
  Thrombosis will be assessed clinically and confirmed by ultrasonographic exam

CONTACTS AND LOCATIONS:
Overall Officials: Annabel Blasi, MD, PhD, Principal Investigator — Hospital Clinic Barcelona. IDIBAPS
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Cruces, Bilbao

IPD SHARING:
Plan to Share IPD: Undecided